CLINICAL TRIAL: NCT05761626
Title: Mechanical Power Normalized to Compliance in Patients With Acute Respiratory Distress Syndrome
Brief Title: Mechanical Power Normalized to Compliance in ARDS
Status: Completed | Type: Observational
Sponsor: Ramos Mejía Hospital (Other)
Responsible Party: Principal Investigator, Roberto Santa Cruz, Principal Investigator, Ramos Mejía Hospital
Other Study IDs: Universidad de Magallanes
Record Dates: First submitted 2023-02-20; First posted 2023-03-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with MP/Crs < = 0.48 j/min/ml/cmH2O: Patients with MP/Crs < = 0.48 j/min/ml/cmH2O
  Interventions: Other: MP/Crs assessment < = 0.48 J/min/ml/cmH2O
- Patients with MP/Crs > 0.48 j/min/ml/cmH2O: Patients with MP/Crs > 0.48 j/min/ml/cmH2O

INTERVENTIONS:
Other: MP/Crs assessment < = 0.48 J/min/ml/cmH2O — Assessment of the ventilatory variables according to the MP/Crs value (<= or > 0.48 J/min/ml/cmH2O)
  Groups: Patients with MP/Crs < = 0.48 j/min/ml/cmH2O

SUMMARY:
Mechanical power (MP) is a summary variable, which includes static and dynamic respiratory parameters, is associated with ventilator-induced lung injury. MP is transferred primarily to smaller functional lung size, often referred to as "baby lung" (BL). Functional lung size (BL) is associated with respiratory system compliance (Crs). For this reason, MP normalized to Crs (MP/Crs) could be an important parameter to evaluate. The objectives of this study were to compare variables according to the MP/Crs cut-off point and to identify the MP components associated with MP/Crs.

DETAILED DESCRIPTION:
In patients with acute respiratory distress syndrome (ARDS), undergoing mechanical ventilation (MV), each respiratory cycle transfers a specific amount of mechanical energy to the lung, aimed to expand and overcome airway resistance. The total mechanical energy multiplied by the respiratory rate (RR) defines the mechanical power (MP). It has been hypothesized that a smaller functional lung size, often referred to as "baby lung" (BL), increases mechanical energy transfer that exacerbates lung damage. Functional lung size (BL) is associated with respiratory system compliance (Crs). Whatever the size of this operational BL, protective ventilation strategies should be aimed at preserving its size and functionality, to avoid ventilator-induced lung injury (VILI). For this reason, MP normalized to Crs (MP/Crs) could be an important parameter to evaluate. Preclinical studies have found that VILI arises primarily from a combination of MP components and not from any of its components individually. We believe that MP/Crs should have the same behavior in relation to MP components as a whole. Therefore, the objectives of this study are to compare variables according to the MP/Crs cut-off point and to identify the MP components associated with MP/Crs.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been receiving mechanical ventilation (MV) and have been defined as with ARDS according to the Berlin definition

Exclusion Criteria:

* patients with chronic pulmonary disease
* patients with an expected duration of MV shorter than 48 h
* patients with a high risk of death within 3 months for reasons other than ARDS
* patients having made the decision to withhold life-sustaining treatment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been receiving mechanical ventilation (MV) and have been defined as with ARDS according to the Berlin definition
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
To compare variables according to the MP/Crs (J/min/ml/cmH2O) cut-off point | Third day of mechanical ventilation
  MP/Crs (J/min/ml/cmH2O) will be used to establish the cut-off and compare variables.

SECONDARY OUTCOMES:
Components of MP associated with MP/Crs (J/min/ml/cmH2O) | Third day of mechanical ventilation
  Through a multivariate analysis, the association between MP/Crs (J/min/ml/cmH2O) and the components of MP will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Rio Gallegos, Río Gallegos, Santa Cruz Province, Argentina

IPD SHARING:
Plan to Share IPD: No
The data will be uploaded in an Excel document and shared with all the researchers participating in the study.

REFERENCES:
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Maj R, Palermo P, Gattarello S, Brusatori S, D'Albo R, Zinnato C, Velati M, Romitti F, Busana M, Wieditz J, Herrmann P, Moerer O, Quintel M, Meissner K, Sanderson B, Chiumello D, Marini JJ, Camporota L, Gattinoni L. Ventilatory ratio, dead space, and venous admixture in patients with acute respiratory distress syndrome. Br J Anaesth. 2023 Mar;130(3):360-367. doi: 10.1016/j.bja.2022.10.035. Epub 2022 Dec 2. PMID 36470747
- [Background] Marini JJ, Jaber S. Dynamic predictors of VILI risk: beyond the driving pressure. Intensive Care Med. 2016 Oct;42(10):1597-1600. doi: 10.1007/s00134-016-4534-x. Epub 2016 Sep 16. No abstract available. PMID 27637717
- [Background] Marini JJ. How I optimize power to avoid VILI. Crit Care. 2019 Oct 21;23(1):326. doi: 10.1186/s13054-019-2638-8. No abstract available. PMID 31639025
- [Background] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Background] Sinha P, Fauvel NJ, Singh S, Soni N. Ventilatory ratio: a simple bedside measure of ventilation. Br J Anaesth. 2009 May;102(5):692-7. doi: 10.1093/bja/aep054. Epub 2009 Apr 3. PMID 19346233
- [Background] Sinha P, Calfee CS, Beitler JR, Soni N, Ho K, Matthay MA, Kallet RH. Physiologic Analysis and Clinical Performance of the Ventilatory Ratio in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2019 Feb 1;199(3):333-341. doi: 10.1164/rccm.201804-0692OC. PMID 30211618
- [Background] Urner M, Juni P, Hansen B, Wettstein MS, Ferguson ND, Fan E. Time-varying intensity of mechanical ventilation and mortality in patients with acute respiratory failure: a registry-based, prospective cohort study. Lancet Respir Med. 2020 Sep;8(9):905-913. doi: 10.1016/S2213-2600(20)30325-8. Epub 2020 Jul 28. PMID 32735841
- [Background] Zhang Z, Zheng B, Liu N, Ge H, Hong Y. Mechanical power normalized to predicted body weight as a predictor of mortality in patients with acute respiratory distress syndrome. Intensive Care Med. 2019 Jun;45(6):856-864. doi: 10.1007/s00134-019-05627-9. Epub 2019 May 6. PMID 31062050